CLINICAL TRIAL: NCT02192788
Title: Phase II Study of SBRT as Treatment for Oligometastases in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo de Investigación Clínica en Oncología Radioterapia (Other)
Responsible Party: Principal Investigator, Antonio J Conde Moreno, MD, Grupo de Investigación Clínica en Oncología Radioterapia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBRT-SG 05
Record Dates: First submitted 2014-07-03; First posted 2014-07-17 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Oligometastatic Prostate Cancer
Keywords: SBRT; Oligometastases; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SBRT (Experimental): Stereotactic Body Radiation Therapy for Oligometastases (SBRT)
  Interventions: Radiation: Stereotactic Body Radiation Therapy for Oligometastases

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy for Oligometastases

SUMMARY:
This study aims to probe the effect of SBRT as a treatment oligometastases of prostate cancer, regardless of basal treatment received, and I know the response, biochemical control, the progression-free survival as well as their impact on quality of life.

Primary Objective: Local and symptomatic oligometastases Control of prostate cancer treated by SBRT.

Secondary Objectives: Analyzing biochemical progression rates, progression-free survival, chemotherapy-free survival and overall survival. Analyze toxicities and quality of life of patients before and after treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed prostate cancer, who are currently being oligometastases / oligorrecurrencia after primary treatment for their disease.
* Aged ≥ 18 years
* Time to biochemical recurrence more than 1 year
* PSA doubling time> 3 months
* Less than 5 bone metastases location (including spinal) or lymph node.
* Without other metastases or recurrences by Choline PET or / and NMR Diffusion Length.
* Signed and dated written informed consent form.

Exclusion Criteria:

* Patients currently treatment with abiraterone, enzalutamide, chemotherapy, immunotherapy or radioisotopes.
* Patients unwilling or unable to comply with protocol requirements and scheduled visits.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-08; Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Number of patients without disease progression of prostate cancer treated by SBRT | 5 years
  Number of patients without disease progression of local and symptomatic oligometastases of prostate cancer treated by SBRT expressed as total number and percentage

SECONDARY OUTCOMES:
Overall Survival measured with Kaplan-Meier method | patients will be followed up an average of 5 years
  the time to death will be defined as the time between the date when the patient is treated with SBRT and the date of death, or the last follow-up visit.
Number of patients with an adverse events. | 3 months after the SBRT treatment
  Analyze toxicities in every patient during the first 3 months after the treatment with SBRT. Every significant Adverse Event will be graded as CTC-AE v.4.03. For Pain related adverse events, visual analogic scale (VAS) will be used.
Free disease progression survival measured with Kaplan-Meier method | the patients will be followed up an expected average of 5 years
  the time to disease progression will be defined as the time between the date when the patient is treated with SBRT and the date of biochemical (PSA increased upper to 2 ng/mL) o radiological progression or the last follow-up visit.
Quality of life questionnaire FACT-P | baseline and 3rd month after the SBRT treatment.
  The Functional Assessment Of Cancer Therapy-Prostate Questionnaire (FACT-P) will be performed at baseline and 3 months after the SBRT treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio J Conde Moreno, MD, Principal Investigator — Grupo de Investigación Clínica en Oncología Radioterapia
Locations (22):
- Spain (22):
  - GICOR, Madrid, Las Rozas
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Rey Juan Carlos, Móstoles, Madrid
  - Santa Lucia, Cartagena, Murcia
  - Instituto catalan de Oncología, Barcelona
  - Hospital de Cruces, Bilbao
  - C.H.P. Castellón, Castellon
  - Hospital Dr. Negrin, Las Palmas de Gran Canaria
  - Clínica QUIRON, Madrid
  - Hospital central de la defensa Gomez Ulla, Madrid
  - Hospital de Sanchinarro, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital de Navarra, Navarro
  - Hospital Universitario Clínico de Salamanca, Salamanca
  - Hospital marques de Valdecilla, Santander
  - ERESA H. General de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Do Mexoeiro, Vigo
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Conde-Moreno AJ, Lopez-Campos F, Hervas A, Morillo V, Mendez A, Puertas MDM, Valero-Albarran J, Gomez Iturriaga A, Rico M, Vazquez ML, Samper Ots PM, Perez-Romasanta LA, Pastor J, Ibanez C, Ferrer F, Zapatero A, Garcia-Blanco AS, Rodriguez A, Ferrer C. A Phase II Trial of Stereotactic Body Radiation Therapy and Androgen Deprivation for Oligometastases in Prostate Cancer (SBRT-SG 05). Pract Radiat Oncol. 2024 Sep-Oct;14(5):e344-e352. doi: 10.1016/j.prro.2024.04.022. Epub 2024 Jun 29. PMID 38944806